CLINICAL TRIAL: NCT01347411
Title: Effectiveness of the Treatment With CONTINUOUS POSITIVE AIRWAY PRESSURE (CPAP) in Stable Heart Failure With Ejection Fraction More Than 45% and Sleep Disordered Breathing
Brief Title: Effectiveness of the Treatment With Continuous Positive Airway Pressure(CPAP)in Stable Heart Failure With Ejection Fraction More Than 45% and Sleep Disordered Breathing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Basque Health Service (Other Government)
Responsible Party: Carlos Javier Egea Santaolalla, Hospital Txagorritxu
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DIDAS
Record Dates: First submitted 2011-04-13; First posted 2011-05-04 (Estimated); Last update posted 2011-05-04 (Estimated); Status verified 2011-04

CONDITIONS: Heart Failure; Sleep Respiratory Disorders
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): Usual treatment
- CPAP (Experimental): Treatment with CPAP
  Interventions: Procedure: CPAP

INTERVENTIONS:
Procedure: CPAP — Treatment with CPAP
  Arms: CPAP

SUMMARY:
The respiratory sleep disorders are a major cardiovascular risk factor. In fact there is enough scientific evidence that supports the association between apnea-hypopnea syndrome (SASH) and cardiovascular disease (hypertension, stroke, heart failure ....The objective of this study is to estimate the effectiveness of the continuous positive pressure airway (CPAP) in patient with chronic heart failure with normal ejection fraction but dyastolic dysfunction and sleep disordered breathing during the sleep.

ELIGIBILITY:
Inclusion Criteria:

1. Ejection fraction> 45%, which also ruled out significant left ventricular dilation
2. At least two abnormal indices of diastolic function.

Exclusion Criteria:

1. Not sinus rhytm
2. Severe lung disease (FEV1 or FVC less than 50%)
3. Significant valvular or congenital heart disease, primary
4. Unstable angina, myocardial infarction or cardiac surgery within three months prior to inclusion
5. Hypertrophic Cardiomyopathy
6. Presence of significant psychiatric disorders.
7. Severe Hypersomnia . (Epworth> 20)
8. Severe pulmonary hypertension measured by Doppler,
9. Facial deformity and / or defect of nasal patency.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 420 (Actual)
Dates: Start 2007-09; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
number of patients without diastolic dysfunction | One year
  number of patient without diastolic dysfunction defined by any of this parametres: TRI (isovolumetric relaxation time):> 105 ms (> 50 years),> 100 ms (30-50 years). 2. Wave ratio E / A wave <1 and deceleration time> 220 ms (under 50) and E / A <0.5 and deceleration time> 280 ms (50 +). 3. Relationship between systolic and diastolic wave flow following pulmonary vein (S / D): S / D> 1.5 (under 50) and S / D> 2.5 (over 50). A wave velocity of pulmonary venous flow> 35 cm / s. Flow propagation velocity by color M-mode <45 cm / s. E wave peak velocity by DTI of the ring: Em <5 cm / s
number of hospital admissions for any cause | One year